CLINICAL TRIAL: NCT04665791
Title: A Human Controlled Infection Study to Assess Colonisation and Immunogenicity Following Nasal Inoculation of Malian Adults with Reconstituted Lyophilised Wild Type Neisseria Lactamica (Lactamica Etape 1)
Brief Title: A Human Controlled Infection Study with Neisseria Lactamica in Malian Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Vaccine Development - Mali (Other)
Collaborators: University of Southampton (Other); University of Maryland (Other); University College, London (Other); University of Oxford (Other); Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 62190
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Meningitis, Meningococcal
Keywords: Meningitis; Controlled human infection; Healthy volunteer; Neisseria lactamica; Lyophilization
MeSH Terms: conditions — Meningitis, Meningococcal; Meningitis

STUDY DESIGN:
Intervention Model Description: A prospective dose-ranging human challenge study. Nasal inoculation with reconstituted, previously lyophilised Neisseria lactamica with dose escalation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Challenge (Experimental): Challenge participants will be inoculated intranasally with reconstituted, previously lyophilised Neisseria lactamica (LyoNlac). The initial dose will be 10^5 colony forming units and will be escalated to a maximum of 10^7 colony forming units to find the dose which successfully colonises at least 70% of volunteers.
  Interventions: Biological: Intranasal inoculation with Neisseria lactamica

INTERVENTIONS:
Biological: Intranasal inoculation with Neisseria lactamica — Lyophilised Neisseria lactamica will be reconstituted and administered to participants intranasally.

SUMMARY:
This study is part of a series of projects to improve protection against meningitis. Previously, researchers have given nose drops containing N. lactamica to over 400 volunteers and shown that many of them become colonised with N. lactamica without causing any illness or disease. This has previously been shown to prevent people from becoming colonised with N. meningitidis which can cause meningitis. This study aims to give nose drops containing N. lactamica to healthy adults in Mali, to see if they become safely colonised. In the future the study team would like to find out how N.lactamica helps children resist N.meningitidis, and develop new vaccines that exploit that mechanism.

DETAILED DESCRIPTION:
In this pilot research, the study team will use a methodology of nasal inoculation with reconstituted lyophilised N. lactamica (hereafter LyoNlac) developed in a previous, UK-based, human challenge study. This methodology and will be developed further and validated in healthy Malian adults.

A dose-ranging strategy will be used, starting with the dose identified as the standard inoculum in healthy adults in the UK, which was the dose required to induce colonisation in approximately 80% of volunteers. The dose will be escalated to a dose able to induce a similar level of colonisation in Malian adults. This study will inform the study team whether intranasal inoculation of reconstituted lyophilised Nlac (hereafter, lyoNlac), can result in immunising colonisation of adult Malian volunteers and the optimal dose to achieve this. This dose and methodology will then be used in future studies looking at the duration and immunogenicity of colonisation induced by LyoNlac in Mali.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years inclusive on the day of enrolment residing outside the demographic surveillance area
* Able and willing (in the investigator's opinion) to understand and comply with all study requirements including availability for all study follow up visits
* Provide written informed consent to participate in the trial
* For females only, all the following:
* willingness to practice continuous effective contraception at least until the Day 28 visit is complete
* negative urine pregnancy test on the screening day
* negative urine pregnancy test on inoculation day

Exclusion Criteria:

Eligibility Minimum Age: 18 Years Maximum Age: 45 Years Sex: All Gender Based: No Accepts Healthy Volunteers: Yes

Criteria: Inclusion Criteria:

* Healthy adults aged 18 to 45 years inclusive on the day of enrolment residing outside the demographic surveillance area
* Able and willing (in the investigator's opinion) to understand and comply with all study requirements including availability for all study follow up visits
* Provide written informed consent to participate in the trial
* For females only, all the following:
* willingness to practice continuous effective contraception at least until the Day 28 visit is complete
* negative urine pregnancy test on the screening day
* negative urine pregnancy test on inoculation day

Exclusion Criteria:

* N. lactamica detected on throat swab taken at the screening visit
* Individuals who have an ongoing acute illness at the time of inoculation
* Individuals who have been involved in other clinical trials involving receipt of an investigational product over the last 12 weeks or if there is planned use of an investigational product during the study period
* Use of systemic antibiotics within the period 30 days prior to the challenge
* Any confirmed or suspected immunosuppressive or immune-deficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication (including oral steroids) within the past 6 months (topical steroids are allowed)
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* History of allergic disease or reactions to soya.
* Any clinically significant abnormal finding on clinical examination or screening investigations
* History of any surgery to the nose or throat in the previous 3 months
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
* Occupational, household or intimate contact with immunosuppressed persons
* Positive pregnancy test or lactation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Establish the impact of nasal inoculation of healthy Malian volunteers with reconstituted lyophilised Neisseria lactamica by assessing nasopharyngeal colonisation with Neisseria species | 6 months
  Throat swabs will be taken at standardised visits and analysed for nasopharyngeal colonisation with Neisseria species. Standard tests include culture and polymerase chain reaction (PCR)
Establish the effect of the nasal inoculation of healthy Malian volunteers with reconstituted lyophilised Neisseria lactamica by collecting information about symptoms | 6 months
  Information about symptoms will be collected at standardised visits. Any symptoms will be recorded and assessed by a study doctor. If deemed necessary by the study doctor further tests will be requested.
Analyse the haemoglobin of healthy Malian volunteers inoculated with reconstituted lyophilised Neisseria lactamica | 3 months
  Blood samples will be taken at specified time points and compared to those collected at baseline. Any change in results will be recorded and, if deemed necessary by the medical team, further tests will be requested. Standard tests - haemoglobin - g/dL
Analyse the white cell count of healthy Malian volunteers inoculated with reconstituted lyophilised Neisseria lactamica | 3 months
  Blood samples will be taken at specified time points and compared to those collected at baseline. Any change in results will be recorded and, if deemed necessary by the medical team, further tests will be requested. Standard tests - white cell count - x 10^9/L
Analyse the platelet count of healthy Malian volunteers inoculated with reconstituted lyophilised Neisseria lactamica | 3 months
  Blood samples will be taken at specified time points and compared to those collected at baseline. Any change in results will be recorded and, if deemed necessary by the medical team, further tests will be requested. Standard tests - Platelet count x 10^9/L
Analyse the biochemistry blood results (ALT) of healthy Malian volunteers inoculated with reconstituted lyophilised Neisseria lactamica | 3 months
  Blood samples will be taken at specified time points and compared to those collected at baseline. Any change in results will be recorded and, if deemed necessary by the medical team, further tests will be requested. Standard tests - ALT
Analyse the biochemistry blood results (Creatinine) of healthy Malian volunteers inoculated with reconstituted lyophilised Neisseria lactamica | 3 months
  Blood samples will be taken at specified time points and compared to those collected at baseline. Any change in results will be recorded and, if deemed necessary by the medical team, further tests will be requested. Standard tests - Creatinine (mg/dL)

SECONDARY OUTCOMES:
The dose of reconstituted lyophilised Neisseria lactamica required for nasopharyngeal colonisation in at least 70% of inoculees | 6 months
  The dose will be confirmed by throat swabs taken from participants and analysed for bacteria by culture and polymerase chain reaction. The desired dose will be confirmed when at least 70%o of inoculees are colonised
To measure Neisseria lactamica specific immunity following nasal inoculation with reconstituted lyophilised Neisseria lactamica | 1 year
  Blood samples will be collected at standardised visits and antibody levels (mg/dL) will be measured to assess if those colonised with Neisseria lactamica show an increase in antibody levels in comparison to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Read, MD FRCP, Principal Investigator — University of Southampton; Samba Sow, MD, Principal Investigator — Center for Vaccine Development - Mali; Milagritos Tapia, MD, Principal Investigator — University of Maryland
Locations (1):
- CVD Mali, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gbesemete DF, Haidara F, Laver JR, Ibrahim M, MacLennan J, Dale AP, Gorringe AR, Traore Y, Diallo F, Badji H, Traore A, Onwuchekwa U, Jones E, Webb C, Guy J, Theodosiou AA, Faust SN, Sow SO, Heyderman RS, Tapia MD, Read RC. Controlled Human Infection of Healthy Adults With Lyophilized Neisseria lactamica Induces Asymptomatic, Immunogenic Nasopharyngeal Carriage in the United Kingdom and Mali. Open Forum Infect Dis. 2026 Jan 7;13(1):ofaf809. doi: 10.1093/ofid/ofaf809. eCollection 2026 Jan. PMID 41574175